CLINICAL TRIAL: NCT05846256
Title: Evaluation of Single and Double DNA Strand Breaks in Males With Unexplained Infertility Attending Fertility Treatment
Brief Title: Single and Double DNA Strand Breaks in Males With Unexplained Infertility Attending Fertility Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peter Humaidan (Other)
Collaborators: ExamenLab Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Consultant, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Other Study IDs: Doublestrand DNA Fragmentation
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Infertility, Male
Keywords: Sperm DNA Fragmentation; Lifestyle; Doublestrand DNA Fragmentatio
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infertile male: Men with unexplained infertility
  Interventions: Other: Sperm DNA Fragmentation
- Donors (control): Fertile sperm donors
  Interventions: Other: Sperm DNA Fragmentation

INTERVENTIONS:
Other: Sperm DNA Fragmentation — Sperm DNA Fragmentation analysis.

SUMMARY:
The aim of this study is to investigate the extent of double-stranded DNA damage in sperm in men with unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertile men who will undergo 1st or 2nd IVF treatment
* Age over 18 years
* Normal sperm parameters according to WHO criteria
* IVF treatment

Exclusion Criteria:

- ICSI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with unexplanied infertility undergoing fertility treatment
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of double-stranded DNA damage in sperm of men with unexplained infertility. | 30-60 minutes
  Sperm DNA Fragmentation done with a Comet Assay analysis

SECONDARY OUTCOMES:
The proportion of single-stranded DNA damage in sperm of men with unexplained infertility | 30-60 minutes
  Sperm DNA Fragmentation done with a Comet Assay analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic Regional Hospital Skive, Skive, Denmark

IPD SHARING:
Plan to Share IPD: No